CLINICAL TRIAL: NCT06260462
Title: Conventional Glucocorticoids vs. Dual-release Hydrocortisone Effects on Metabolic, Cardiovascular, and Bone Outcomes in Treatment-naïve Patients With Adrenal Insufficiency: a 10-year Prospective Randomised Study
Brief Title: Effects of Steroid Replacement Therapy on Metabolic, Cardiovascular and Bone Outcomes in Adrenal Insufficiency
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Palermo (Other)
Responsible Party: Principal Investigator, Carla Giordano, professor, University of Palermo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10 years adrenal insufficiency
Record Dates: First submitted 2024-01-24; First posted 2024-02-15 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Adrenal Insufficiency
MeSH Terms: conditions — Adrenal Insufficiency | interventions — Hydrocortisone; Cortisone

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional steroid treatment (Experimental): Cortisone acetate and hydorocortisone will be administered in two daily doses
  Interventions: Drug: Conventional glucocortidois
- Dual-release hydrocortisone (Experimental): Dual-release hydrocortisone will be administered once daily
  Interventions: Drug: dual-release hydrocortisone

INTERVENTIONS:
Drug: dual-release hydrocortisone — Oral tablets 20-25-30-40 mg/day
  Other Names: Plenadren
  Arms: Dual-release hydrocortisone
Drug: Conventional glucocortidois — Oral tablets 10-15-20-25-37,5-50-62,5 mg/day
  Other Names: hydrocortisone; cortisone acetate
  Arms: Conventional steroid treatment

SUMMARY:
The current study is a randomized, open study aimed to compare the effects of conventional glucocorticoid replacement treatment and dual-release hydrocortisone on anthropometric, metabolic, cardiovascular and bone outcomes in treatment-naïve patients with primary adrenal insufficiency and secondary adrenal insufficiency in a 10 year-observation period.

DETAILED DESCRIPTION:
Adrenal insufficiency (AI) can be caused by a disease involving the adrenal gland resulting in inadequate secretion of adrenal cortex hormones, primary adrenal insufficiency (PAI). Secondary adrenal insufficiency (SAI) results from a decreased level of adrenocorticotrophin hormone (ACTH) released from the pituitary gland.

The mainstay of treatment of PAI and SAI is glucocorticoid (GC) replacement therapy. Conventional steroid replacement therapy includes cortisone acetate and hydrocortisone administered 2-3 times a day with the highest dose in the morning and the lowest dose in the afternoon. These dosing regimens have been designed to mimic the peak of cortisol secretion in the morning and avoid overdosing during the night hours, even though a higher risk of developing comorbidities has been shown, notably in patients treated with higher evening doses.

In patients with AI on conventional steroid replacement therapy, mortality remains higher than in the general population, mainly due to non-physiological daily GC overexposure and to inadequate cortisol exposure during stress-related events and illness.

Studies aiming to evaluate the long-term clinical outcomes of patients with AI on conventional steroid replacement therapy clearly showed increased comorbidities, mainly related to the dose used.

By contrast, dual-release hydrocortisone (DR-HC) is characterized by once-daily administration with high release of hydrocortisone immediately after intake and a very low release in the evening and nocturnal hours. The switch from conventional GC therapy to DR-HC has been shown to be associated with improvement in BMI, hepatic, bone and glucometabolic parameters and QoL. However, long-term clinical outcomes of patients treated with DR-HC in patients naïve to steroid treatment are not known.

ELIGIBILITY:
Inclusion Criteria:

* Adrenal insufficiency

Exclusion Criteria:

* Exclusion criteria were adrenocortical carcinoma and congenital adrenal hyperplasia

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2012-01-01 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Change of body weight | 0, 5 years, 10 years
  Single outcome measurement of body weight (kg).

SECONDARY OUTCOMES:
Change of anthropometric parameters | 0, 5 years and 10 years
  waist circumference
Change of metabolic parameters | 0, 5 years and 10 years
  Composite outcome including evaluation of total cholesterol, HDL cholesterol, LDL cholesterol and triglycerides, HbA1c and fasting blood glucose
Change of insulin sensitivity parameters | 0, 5 years and 10 years
  the Isi-Matsuda index
Change of cardiovascular parameters | 0, 5 years and 10 years
  Measurement of interventricular septum at diastole (IVSd) and the thickness of the posterior wall (PWT) by high-resolution M-B-mode transthoracic echocardiography
Change of bone metabolic parameters | 0, 5 years and 10 years
  Composite outcome including calcium, phosphorus, Vitamin D, PTH, creatinine (all measured in mg/dL)
Change of bone density | 0, 5 years and 10 years
  Bone mineral density quantified by Dual X-Ray Absorptiometry (DEXA)
Change of vascular parameters | 0, 5 years and 10 years
  Measurement carotid intima media thickness by high-resolution M-B-mode echography

IPD SHARING:
Plan to Share IPD: Yes
Study protocol could be available on request
Supporting Information: Study Protocol
Time Frame: 2 years
Access Criteria: Send an email to carla.giordano@unipa.it

REFERENCES:
- [Derived] Guarnotta V, Di Stefano C, Tomasello L, Maniscalco L, Pizzolanti G, Arnaldi G, Giordano C. Conventional steroids vs. dual-release hydrocortisone on metabolic, cardiovascular, and bone outcomes in adrenal insufficiency: a 10-year study. Eur J Endocrinol. 2024 Aug 30;191(3):300-311. doi: 10.1093/ejendo/lvae107. PMID 39171906